CLINICAL TRIAL: NCT05024903
Title: A Randomized Trial of a Novel E-health Platform (Plan Well GuideTM)
Brief Title: A Novel E-health Platform
Acronym: PWG
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to enroll enough patients in the time allotted. Study deemed infeasible.Dece
Sponsor: Daren K. Heyland (Other)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Director of Clinical Evaluation Research Unit, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: PWG
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Aging Well; Decision Making; Illness, Critical
MeSH Terms: conditions — Critical Illness | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: (PWG 1.0) (Active Comparator): Those randomized to PWG 1.0 would have already completed their serious illness medical planning. Further involvement in the trial will be solely for the purposes of the outcome data collection
  Interventions: Other: Standard of care
- Intervention group: PWG 2.0 (Active Comparator): Serious illness medical planning plus the novel e-health platform designed to help people more broadly think and plan ahead
  Interventions: Other: Serious illness medical planning plus the novel e-health platform (PWG 2.0)

INTERVENTIONS:
Other: Serious illness medical planning plus the novel e-health platform (PWG 2.0) — PWG 2.0 consists of the following components:
  1. A diagnostic questionnaire, "Preparedness for the Future Questionnaire" and bench-marked report that helps users assess their strengths, weaknesses and opportunities for improvement.
  2. A comprehensive e-workbook that helps users understand the science behind personal behavior change.
  3. Links to webpages with additional e-workbooks and curated content aimed to help users progress on the 30 different attitudes, behaviors, and activities that portend for a better future (topics listed in Appendix A).
  4. E-messages delivered via emails (via text an option for those that prefer) with tailored content designed to provide multiple nudges to guide the user to progress through our content.
  5. Monthly newsletter with current topics and issues related to the 30 topics and behavior change in general.
  6. A virtual consultation with Dr. Heyland, creator of PWG and principal investigator.
  Arms: Intervention group: PWG 2.0
Other: Standard of care — Participants are not planning for their future (PWG 2.0) or using the e-health platform
  Arms: Control Group: (PWG 1.0)

SUMMARY:
The purpose of the current trial is to evaluate a novel e-health platform. Overall Hypothesis: Participants who receive Plan Well Guide (PWG) 2.0 will make more progress in their 'preparations' as measured by "Preparedness for the Future Questionnaire (PREP FQ)" at 6 months and, consequently, experience greater improvements in their psychological well-being (PWB), health status, and life satisfaction at 12 months compared to participants receiving PWG 1.0 (Advance Serious Illness module only). Study Design: The investigators propose to conduct a multi-site randomized trial to evaluate a novel e-health platform. Overall Hypothesis: Participants who receive Plan Well Guide (PWG) 2.0 will make more progress in their 'preparations' as measured by "Preparedness for the Future Questionnaire (PREP FQ)" at 6 months and, consequently, experience greater improvements in their psychological well-being (PWB), health status, and life satisfaction at 12 months compared to participants receiving PWG 1.0 (Advance Serious Illness module only).Study Design: We propose to conduct a multi-site randomized trial. Setting: Several sites in Lethbridge Alberta. a sample of primary care clinics as well as recruit online participants. Study Population: The investigators plan to include interested participants that are aged between 25 to 70 years of age. We will exclude participants that don't speak English or do not have internet access/email addresses, and already have a high PWB score. Study Intervention: Eligible participants will then be randomly allocated to 2 groups: PWG 1.0 or PWG 2.0.Outcomes: The primary outcome for this trial will be an overall score of PWB questionnaire; key secondary outcomes include PWB domain scores, SF-12,single-item rating of life satisfaction, all measured at 6 and 12 months. Additional outcomes include 'days off work' and health care utilization. Significance: This study will be the first large multi-centre trial examining the effects of a novel e-health platform aimed at improving people's psychological well-being and health status as well as their preparedness for serious illness decision-making during this time of a global pandemic. Results of this trial will likely affect the state of preparedness of individuals, and if wide disseminated, may have a dramatic effect on the health and well-being of a broad segment of the population.

ELIGIBILITY:
Inclusion Criteria:

* 25-70 years old

Exclusion Criteria:

* don't speak or read English
* no home internet access
* a baseline PWB score of 4.5 or greater

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Overall Preparedness for the Future Question score | 6 months
  All scores were re-scaled to range between 0 (worst -lowest possible total points given the applica- ble answered questions) and 100 (best -highest possible total points given applicable answered questions).
  Measured for the Phase II trial: the questionnaire contains 34 items in 8 distinct domains ("Medico-legal", "Social", "Psychological Well-being", "Planning", "Enrichment", "Positive Health Behaviors", "Negative Health Behaviors", and "Late-life Planning")
Item scores for Preparedness for the Future Question score | 6 months
  Measured for the Phase II trial

OTHER OUTCOMES:
Overall score of Psychological Well Being Scale | 12 months
  Scale is 42 to 294 and the higher scores indicate greater wellbeing

CONTACTS AND LOCATIONS:
Locations (1):
- City of Lethbridge, Lethbridge, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howard M, Elston D, Borhan S, Hafid A, Arora N, Forbes R, Bernard C, Heyland DK. Randomised trial of a serious illness decision aid (Plan Well Guide) for patients and their substitute decision-makers to improve engagement in advance care planning. BMJ Support Palliat Care. 2022 Mar;12(1):99-106. doi: 10.1136/bmjspcare-2021-003040. Epub 2021 Jun 30. PMID 34193434
- [Background] Heyland DK, Heyland R, Bailey A, Howard M. A novel decision aid to help plan for serious illness: a multisite randomized trial. CMAJ Open. 2020 Apr 28;8(2):E289-E296. doi: 10.9778/cmajo.20190179. Print 2020 Apr-Jun. PMID 32345707
- [Background] Howard M, Slaven M, Bernard C, Borhan S, Elston D, Arora N, Tan A, Heyland DK. Decision support intervention (Plan Well Guide) for patients and their substitute decision-makers to improve engagement in advance care planning: protocol for a randomised trial. BMJ Open. 2019 Sep 20;9(9):e027897. doi: 10.1136/bmjopen-2018-027897. PMID 31542737
- [Background] Heyland DK, Pope JP, Jiang X, Day AG. Determining the psychometric properties of a novel questionnaire to measure "preparedness for the future" (Prep FQ). Health Qual Life Outcomes. 2021 Apr 15;19(1):122. doi: 10.1186/s12955-021-01759-z. PMID 33858414